CLINICAL TRIAL: NCT05030168
Title: The Effects of Low Protein Diet Supplemented With Ketoanalogues on Preservation of Residual Kidney Function Among Patients Undergoing Incremental Dialysis
Brief Title: Effects of Low Protein Diet Supplemented With Ketoanalogues on Preservation of Kidney Function in Incremental Dialysis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Kearkiat Praditpornsilpa, Professor of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB NO.779/62
Record Dates: First submitted 2020-10-12; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Kidney Function; Hemodialysis
MeSH Terms: interventions — ketosteril; Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (No Intervention): Twice weekly hemodialysis program plus regular protein diet (1.0 g/kg/day) every day
- Ketosteril (Experimental): Incremental hemodialysis program, starting from once weekly hemodialysis/hemodialysis filtration(HDF) plus low protein diet (0.6 g/kg/day) and ketoanologues 0.12g/kg/day supplementation on non-dialysis days and regular protein diet (1.0-1.2 g/kg/day) on dialysis day
  Interventions: Drug: Ketosteril

INTERVENTIONS:
Drug: Ketosteril — ketoanalogues of essential amino acid
  Other Names: incremental hemodialysis; low protein diet
  Arms: Ketosteril

SUMMARY:
The investigators hypothesized that combination of incremental hemodialysis and ketoanologues will better preserve residual kidney function and maintenance of nutritional status among the incident ESRD patients during the early initiation of chronic dialysis. This hypothesis has been a new concept of chronic hemodialysis initiation for End stage renal disease (ESRD) patients

DETAILED DESCRIPTION:
The investigators plan to conduct the first randomized Phase IIA clinical trial to investigate the efficacy of incremental hemodialysis and moderately low protein diet combined with ketoanologues supplementation on preservation of residual kidney function, inflammatory status and nutritional parameters among incident chronic dialysis patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at screening
* Stable CKD stage 5 not yet on dialysis with residual kidney function 5-10 ml/min/1.73m2 by CKD-EPI equation
* Urine output ≥ 800 ml/day
* Willing to participate in the study and can provide inform consent

Exclusion Criteria:

* Rapid glomerular filtration rate (GFR) progression defined as a decline of eGFR >10 ml/min/1.73m2 by CKD-EPI equation in the prior 6 months before enrollment
* Presence of wasting diseases, cancer cachexia, tuberculosis, AIDS wasting syndrome
* Other active infection/inflammation determined by CRP >10 mg/L
* Severe gastrointestinal problem: persistent nausea/vomiting, dysphagia, chronic diarrhea, severe malabsorption
* Conditions at baseline requiring withdrawal from the study including severe protein energy wasting by SGA and MIS score, prior kidney transplantation with immunosuppressive agents or other serious medical conditions.
* Pregnancy
* Uncontrolled hypercalcemia (persistent serum Ca ≥10.5 mg/dl)
* BMI ≥ 35 kg/m2
* Hypersensitivity to the active substances or to any of the excipients of Ketosteril
* Disturbed amino acid metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
residual renal function | 12 months
  To demonstrate superiority effect of incremental hemodialysis (HD) protocol (initiate with once-weekly hemodialysis) plus ketoanalogues-supplemented low-protein diet during non-dialysis days over the standard HD protocol (initiate with twice weekly hemodialysis) on preservation of residual renal function (renal urea clearance) at 12 months.

SECONDARY OUTCOMES:
visceral protein | 12 months
  To compare serum albumin levels between the two treatment groups over 12 months.
structural protein | 12 months
  To compare muscle mass between the two treatment groups over 12 months.
muscle function | 12 months
  To compare muscle strength between the two treatment groups over 12 months.

IPD SHARING:
Plan to Share IPD: No